CLINICAL TRIAL: NCT05415878
Title: Improving Diabetic Foot Ulcer Offloading: A Pilot Study on the Impact of Removable Cast Walker Design Factors on Usability
Brief Title: Impact of Removable Cast Walker Design on Usability for Patients With Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Noah Rosenblatt, Associate Professor, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK131303
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tall RCW (Other)
  Interventions: Device: RCW design form
- Short RCW with contralateral lift (Other)
  Interventions: Device: RCW design form

INTERVENTIONS:
Device: RCW design form — Tall RCW= a knee high removable cast walker with an offloading insole
  Short RCW= an ankle high (extending up the leg just past the ankle) removable cast walker with an offloading insole, paired with an external shoe lift to be used with a diabetic shoe on the contralateral limb

SUMMARY:
Within their lifetime, over 30% of people living with diabetes will develop a diabetic foot ulcer (DFU), many of which will never heal and may require amputation. Removable cast walkers (RCWs) are commonly prescribed to offload (treat) DFUs. While RCWs are prescribed to be worn during all weight bearing activities, adherence to this prescription is low. This is a serious concern given that low adherence predicts poor DFU healing. This study will provide pilot/feasibility data to inform a larger clinical trial to evaluate the impact of existing RCW designs on adherence and DFU healing. We will also quantify the effect of RCW form on biomechanical and self-reported measures related to usability. Our working hypothesis is that healing outcomes with a given RCW will be predicted by biomechanical and self-reported measures of RCW usability, with the predictive relationship partly explained by the effect of these measures on adherence.

ELIGIBILITY:
Inclusion Criteria:

* presence of a full thickness plantar (forefoot) diabetic foot ulcer ≥1cm2 that is being treated on an outpatient basis with a University of Texas wound classification of 1A-C or 2 A-C;
* self-reported ability to walk for at least two continuous minutes at a self-selected speed
* confirmation of the presence of diabetic peripheral neuropathy as identified by failure to detect a 10 gram Semmes Weinstein Monofilament on either foot at one of four sites tested (1st, 3rd, 5th metatarsal heads, and plantar surface of hallux) OR a vibration perception threshold value of 25 or more at either hallux.

Exclusion Criteria:

* lower extremity amputation more proximal than transmetatarsal on either limb
* chronic kidney disease stage 4 or higher (i.e., currently undergoing dialysis or eGFR<30 within last 60 days)
* active Charcot neuroarthropathy
* severe peripheral arterial disease (non-palpable pulse at posterior tibia and dorsalis pedis arteries, and an ankle brachial index<0.7)
* gait/balance disturbance not attributable to diabetes (e.g. neuromuscular disease or cerebrovascular vascular accident)
* current or previous (within past year) use of an ankle-high RCW or of a contralateral lift to offset an RCW-induced LLD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Offloading adherence | days 0-28
  Percent of weight bearing activity completed while wearing the RCW

SECONDARY OUTCOMES:
Diabetic Foot Ulcer Healing | each clinical visit during days 0-28
  Planimetric wound area
Cumulative plantar tissue stress | days 0-28
  A measure to account for the interaction between offloading capacity of the RCW and device use

OTHER OUTCOMES:
Stability | follow up visit (32-38 days after baseline)
  three separate measures taken during walking and standing (local divergence exponent of he trunk; motor equivalent index during small standing perturbations; and posterior stepping threshold for large perturbations while standing)
Correlates of joint pain | follow up visit (32-38 days after baseline)
  Four separate biomechanical measures related to back, hip and knee pain taken during walking in a motion capture lab (peak pelvic obliquity; peak pelvic tilt; ground reaction force transience; and rate of grand reaction force loading)

CONTACTS AND LOCATIONS:
Overall Officials: Noah J Rosenblatt, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science